CLINICAL TRIAL: NCT05890521
Title: Multi-center Safety Observation of COVID19 Vaccine in a Large Population
Brief Title: Safety Study of COVID19 Vaccine on the Market
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Anhui Zhifei Longcom Biologic Pharmacy Co., Ltd. (Industry)
Collaborators: Hunan Provincial Center for Disease Control and Prevention (Other); Guizhou Center for Disease Control and Prevention (Other); Hainan Center for Disease Control & Prevention (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: LKM-2022-NCV-PM01
Record Dates: First submitted 2022-03-28; First posted 2023-06-06 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: COVID-19
Keywords: Recombinant Novel Coronavirus Vaccine
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Subjects who have not received any Novel Coronavirus vaccine or the full dose of recombinant Novel Coronavirus protein vaccine (CHO cells) shall receive 3 doses of the experimental vaccine intramuscular in the deltoid muscle of the upper arm or complete the remaining doses of the experimental vaccine as per the vaccination schedule at 0, 1, and 2 months, with a dose of 0.5ml for each person.
  Immunized subjects: intramuscular injection of one dose of the experimental vaccine into the deltoid muscle of the upper arm, 0.5ml for each person.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Population Ⅰ (Experimental)
  Interventions: Biological: Recombinant new coronavirus vaccine (CHO cell)

INTERVENTIONS:
Biological: Recombinant new coronavirus vaccine (CHO cell) — Subjects who have not received any Novel Coronavirus vaccine or the full dose of recombinant Novel Coronavirus protein vaccine (CHO cells) shall receive 3 doses of the experimental vaccine intramuscular in the deltoid muscle of the upper arm or complete the remaining doses of the experimental vaccine as per the vaccination schedule at 0, 1, and 2 months, with a dose of 0.5ml for each person.
  Immunized subjects: intramuscular injection of one dose of the experimental vaccine into the deltoid muscle of the upper arm, 0.5ml for each person.

SUMMARY:
Popular topic:Multi-center safety observation of recombinant Novel Coronavirus protein vaccine (CHO cells) in a large population Study population:People aged 18 and above

DETAILED DESCRIPTION:
Overall design:The aim of this study is to carry out safety studies in the large scale healthy population and special population of recombinant New Coronavirus protein vaccine (CHO cell) in China. It will be included in 100 thousand subjects, including 20 thousand special populations. It is planned to enroll 50000 cases in Hunan (including no less than 10000 special people), 40000 cases in Guizhou (including no less than 8000 special people), and 10000 cases in Hainan (including no less than 2000 special people).

Special groups include but are not limited to obesity, chronic metabolic diseases, chronic lung diseases, chronic cardiovascular diseases, tumors, acquired immunodeficiency syndrome, chronic kidney disease, etc. If the researcher determines that it is necessary, the special population shall provide the medical diagnosis certificate or the drug prescription certificate issued by the doctor.

Immunization program: Subjects who have not received any Novel Coronavirus vaccine or the full dose of recombinant Novel Coronavirus protein vaccine (CHO cells) shall receive 3 doses of the experimental vaccine intramuscular in the deltoid muscle of the upper arm or complete the remaining doses of the experimental vaccine as per the vaccination schedule at 0, 1, and 2 months, with a dose of 0.5ml for each person.

Immunized subjects: intramuscular injection of one dose of the experimental vaccine into the deltoid muscle of the upper arm, 0.5ml for each person.

Follow up and record:

1. Passive monitoring:

   After all subjects have been vaccinated, the researcher shall conduct safety education and issue contact cards to the subjects, so that the subjects can contact the researcher in time in case of any discomfort. The researcher shall timely standardize the treatment and collect the AESI or SAE information of the subjects.
2. Active monitoring:

All subjects installed customized APP or Wechat applet through mobile phones on the first 7 days and 30 days after each dose of vaccination, and 3, 6, 9 and 12 months after the last dose of vaccination, and recorded and collected the occurrence of adverse events: ① the first dose of vaccination - 30 days after the whole dose of vaccination, and 30 days after the enhanced vaccination, including the occurrence of all adverse events, including solicited AE (vaccination site (local adverse events) Non inoculated sites (systemic adverse events)) and non solicited AEs; ② First dose - SAE, AESI and pregnancy events within 12 months after full vaccination and 12 months after booster immunization.

The solicitation AE is:

Adverse events at the inoculation site (local): pain, pruritus, erythema, swelling, rash and induration; Non inoculated site (systemic) adverse events: fever, headache, fatigue / fatigue, diarrhea, nausea, vomiting, muscle pain (non inoculated site), acute allergic reaction and cough.

Safety assessment:

AE, AESI and SAE:

1. Collect adverse events of special concern (AESI) from the first dose of vaccination to one year after the whole course of vaccination and one year after intensive immunization, including myocarditis / pericarditis, thrombosis, thrombocytopenia, immune related diseases (psoriasis, rheumatoid arthritis, etc.), nervous system related diseases (glibali syndrome, peripheral neuropathy, bell facial paralysis);
2. Collect serious adverse events (SAE) from the first dose of vaccination to 1 year after the whole course of vaccination and 1 year after intensive immunization;
3. Collect all AEs from the first dose to 30 days after the whole course of vaccination and 30 days after booster immunization.

Pregnancy events:

The pregnancy events from the first dose of vaccination to one year after the whole course of vaccination and one year after the booster vaccination were collected (at the same time, the safety and pregnancy outcome of pregnant women's accidental vaccination were analyzed).

ADE/ VED risk monitoring:

After vaccination (at least one dose of test vaccine) (at each visit), remind the subjects to contact the investigator in time for fever and / or respiratory symptoms (such as dyspnea, sore throat, etc.) and covid-19 suspected or confirmed cases during the study. If the subject is suspected or confirmed to be infected with SARS-COV-2 during the test, he must go to the local Xinguan designated hospital for hospitalization diagnosis and treatment. For confirmed cases, detailed case investigation shall be carried out. In case of aggregated new coronavirus infection or severe, critical and death cases after sars-cov-2 infection during the trial, special investigation shall be carried out. According to the analysis of special investigation results, if there is ADE/ VED phenomenon, an expert meeting shall be held to evaluate whether there is ADE / VED risk.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy people or special people aged 18 and above who meet the requirements of national new coronavirus vaccination (including but not limited to obesity (BMI ≥ 28kg/ m²). Chronic metabolic diseases, chronic lung diseases, chronic cardiovascular diseases, tumors, acquired immunodeficiency syndrome, chronic kidney disease, etc.); If the researcher determines that it is necessary, the special population shall provide relevant written diagnosis certificates, records or drug prescription certificates issued by doctors;
2. The subjects voluntarily participated in the study, signed the informed consent, understood and complied with the requirements of the clinical trial scheme, and were able to understand the research procedures.

Exclusion Criteria:

1. Patients with uncontrolled lymphoproliferative diseases, unresponsive aplastic anemia, active primary immune thrombocytopenia (ITP), uncontrolled bleeding and coagulation diseases, etc;
2. People with uncontrolled epilepsy and other serious neurological diseases (such as transverse myelitis, Guillain Barre syndrome, demyelinating disease, etc.);
3. Patients suffering from acute disease, or acute attack of chronic disease, or uncontrolled severe chronic disease;
4. Previous history of severe allergy to any vaccine or any component of the test vaccine, including aluminum preparation, such as anaphylactic shock, allergic laryngeal edema, Henoch Schonlein purpura, thrombocytopenic purpura, dyspnea, angioneuroedema, etc;
5. The researchers believe that the subject has any disease or condition that may put the subject at unacceptable risk; The subjects could not meet the protocol requirements; Interference with the evaluation of vaccine response.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100000 (Estimated)
Dates: Start 2022-04-02 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
SAE | The period from receipt of the first dose of vaccine to 1 year after receipt of the last dose
  Serious adverse events (SAE) were collected from the first dose to 1 year after full vaccination and 1 year after booster immunization.
AE | The period from receipt of the first dose of vaccine to 1 year after receipt of the last dose
  All AE from the first dose to 30 days after full vaccination and 30 days after booster immunization were collected.
AESI | The period from receipt of the first dose of vaccine to 1 year after receipt of the last dose
  Adverse events of special Interest (AESI) analysis 12 months after first dose-full dose and 12 months after booster dose: incidence of adverse events of special interest

SECONDARY OUTCOMES:
ADE/VED | The period from receipt of the first dose of vaccine to 1 year after receipt of the last dose
  After vaccination (at least one dose of test vaccine) (at each visit), remind the subjects to contact the investigator in time for fever and / or respiratory symptoms (such as dyspnea, sore throat, etc.) and covid-19 suspected or confirmed cases during the study. If the subject is suspected or confirmed to be infected with sars-cov-2 during the test, he must go to the local Xinguan designated hospital for hospitalization diagnosis and treatment. For confirmed cases, detailed case investigation shall be carried out. In case of aggregated new coronavirus infection or severe, critical and death cases after sars-cov-2 infection during the trial, special investigation shall be carried out. According to the analysis of special investigation results, if there is ADE / VED phenomenon, an expert meeting shall be held to evaluate whether there is ADD/ VED risk.

CONTACTS AND LOCATIONS:
Overall Officials: Lidong Gao, Study Chair — Hunan Provincial Center for Disease Control and Prevention
Locations (1):
- Hunan Provincial Center for Disease Control and Prevention, Changsha, Hunan, China